CLINICAL TRIAL: NCT01149148
Title: Effect of Regional Cerebral Oxygen Saturation Monitoring On Neurological Outcome In Patients Undergoing Aortic Arch Surgery
Brief Title: Cerebral Oximetry and Neurological Outcomes in Aortic Arch Surgery Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Wei C Lau, MD, FAHA, M.D., University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: UmichiganHS
Record Dates: First submitted 2010-06-21; First posted 2010-06-23 (Estimated); Results first posted 2012-08-16 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2012-08

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: Aortic Surgeries; Deep Hypothermic Circulatory Arrest
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention INVOS Cerebral Oximetry Monitoring (Active Comparator): Intervention will be initiated if rSO2 drops > 20% from baseline or rSO2 declines below 50%.
  Interventions: Device: INVOS Somanetics Cerebral Oximeter
- Standard of Care (Active Comparator): Blinded cerebral oximetry monitoring with no intervention in surgical procedures and anesthesia without deviation from standard of care.
  Interventions: Device: INVOS Somanetics Cerebral Oximeter

INTERVENTIONS:
Device: INVOS Somanetics Cerebral Oximeter — Sequence of Interventions To Increase Cerebral Oxygen Saturation
  1. Check head and cannula position
  2. Increase mean arterial pressure
  3. Increase pump flow
  4. Increase systemic oxygenation
  5. Increase PaCO2 > 45
  6. Increase anesthetic depth by increasing volatile anesthetic or by administering propofol boluses
  7. Consider PRBC transfusion for Hct < 21%
  Arms: Intervention INVOS Cerebral Oximetry Monitoring
Device: INVOS Somanetics Cerebral Oximeter — INVOS Cerebral Oximetry blinded monitoring with no deviation in surgical procedures or standard of care in anesthesia.
  Arms: Standard of Care

SUMMARY:
The investigators hypothesize that early intervention to optimize regional cerebral oxygenation detected by cerebral oximetry monitoring during deep hypothermic circulatory arrest (DHCA) for patients undergoing aortic surgery will decrease the incidence of transient and permanent neurological dysfunction and improve neurocognitive impairment.

DETAILED DESCRIPTION:
Permanent or transient neurologic dysfunction is a frequent complication in patients undergoing aortic arch surgery.

Two basic methods of brain protection are currently used concomitantly with these complex surgical procedures: deep hypothermic circulatory arrest (DHCA) with or without retrograde cerebral perfusion (RCP)and selective antegrade hypothermic cerebral perfusion. Hypothermic circulatory arrest provides an optimal bloodless operative field, but the incidence of neurological dysfunction increases when the duration of DHCA exceeds 45-50 minutes. Antegrade cerebral perfusion is accomplished by means of direct differential cannulation of the common carotid and right subclavian arteries. Because this technique of brain protection requires a separate perfusion circuit, vigilant monitoring of perfusion pressure and flow rate is of utmost importance. Multiple studies have demonstrated that antegrade selective cerebral perfusion is a well established technique used for cerebral protection during aortic surgery requiring longer periods of DHCA with favorable results in hospital mortality and neurologic outcome. The permanent neurological dysfunction was noted to be 3.8% and the transient neurologic dysfunction to be 7.1% for patients that received antegrade selective cerebral perfusion.

Similarly, neurocognitive studies of DHCA with antegrade cerebral perfusion for patients undergoing aortic arch operations demonstrated 9 % transient neurocognitive impairment for 2 days postoperatively that lasted up to 3 weeks thereafter. Consistent with current surgical practice, the University of Michigan uses antegrade selective cerebral perfusion for all patients undergoing aortic arch surgery requiring DHCA with or without RCP.

A number of monitoring modalities have been used for detecting cerebral malperfusion during aortic surgery or carotid surgery, including transcranial Doppler ultrasound and near infrared spectroscopy (NIRS).

The impact of these monitoring modalities on clinical (neurologic) outcome has not been clearly established. Currently, NIRS has gained considerable attention and acceptance as a non-invasive monitor of cerebral oxygenation. One study showed that a sustained drop in the regional oxygen saturation (rSO2) below 55% for over 5 minutes using cerebral oximetry is closely related to the occurrence of neurological events following aortic surgery. Another study strongly supported that rSO2 should not drop > 20% from baseline to prevent neurologic compromise. In a cohort of elective coronary artery bypass graph (CABG) patients, intervention for cerebral desaturations did show significantly less major organ morbidity or mortality (death, ventilation > 48 h, stroke, myocardial infarction, return for re-exploration. Whether NIRS can be used as a monitor to provide rapid detection and prevention of cerebral ischemia by early intervention that may improve neurological outcome in patients undergoing aortic surgery requiring DHCA with or without RCP is currently unknown.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients 18-80 years of age scheduled for aortic surgery requiring DHCA and intention to use antegrade selective cerebral perfusion with or without RCP

Exclusion Criteria:

* Adult male and female patients 18-80 years of age undergoing aortic surgery NOT scheduled for DHCA
* Patients with ejection fraction < 15%
* Pregnancy
* Prisoners
* Patients mentally impaired (Screening Criteria i.e. MMSE score ≤ 23) History of stroke

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2011-09 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 11-2009 to 9-2011
Groups:
- Intervention INVOS Cerebral Oximetry Monitoring: > 20% drop rSO2 from baseline or declines in rSO2 < 50%
Period: Overall Study
Arm/Group | Intervention INVOS Cerebral Oximetry Monitoring | Standard of Care
Started | 12 | 13
Completed | 10 | 11
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention INVOS Cerebral Oximetry Monitoring | Standard of Care | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 6 | 16
  >=65 years | 2 | 7 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (9.414689) | 62.30769 (11.52088) | 61.44 (10.3846)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Mini Mental State Examination (MMSE)
Description: The Mini-Mental State Examination (MMSE) or Folstein test is a brief 30-point questionnaire test that is used to screen for cognitive impairment. It is also used to estimate the severity of cognitive impairment at a specific time and to follow the course of cognitive changes in an individual over time, thus making it an effective way to document an individual's response to treatment. MMSE = Mini Mental State Exam - measures general orientation and mental status.
  Scores on a scale range from 0 - 30. Scores 23 and below are indicative of problems.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Intervention INVOS Cerebral Oximetry Monitoring | Standard of Care
Number analyzed (Participants) | 12 | 13
scores on a scale | 27 (1.651) | 26.769 (2.048)
Statistical Analysis 1: Comparison: Intervention INVOS Cerebral Oximetry Monitoring vs Standard of Care; The goal was to determine whether cerebral oximetry monitoring during surgery affected cognitive outcomes. Cerebral Oximetry Monitoring unblinded (intervention), and Cerebral Oxymetry Monitoring blinded (control) were given Mini Mental State Exam prior to surgery and three months after surgery. The differences between baseline and 3 month were calculated and compared between the intervention and control groups using t-test; Test type: Superiority or Other; p = 0.678, t-test, 2 sided — A prior threshold for statistical significance is p < 0.05; Mean Difference (Net) = -0.3333, 95% CI 2-sided [-1.36 to 2.02], Standard Deviation 1.626 — The difference between baseline and three months is (baseline - 3 month). The difference in control and intervention is (intervention - control), which in this case is (unblinded - blinded)

2. Primary Outcome: Mini Mental State Examination (MMSE)
Description: as for outcome 1
Time Frame: 3 Months
Population: Not all participants completed 3 month follow up neurocognitive testing.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Intervention INVOS Cerebral Oximetry Monitoring: At the start of surgery two sensor pads will be placed on the patients forehead and attached to the INVOS Monitoring System. If the rSO2 values decrease >20% from baseline or decline below 50 the anesthesiologist will initiate an intervention: Increase mean arterial pressure, check head and cannula position, increase pump flow, increase systemic oxygenation, increase PaCo2 >45, increase anesthetic depth by increaseing volatile anesthetic or administering propoful boluses, consider PRBC transfusion for Hct<21%.
Arm/Group | Intervention INVOS Cerebral Oximetry Monitoring | Standard of Care
Number analyzed (Participants) | 9 | 9
Scores on a scale | 27.667 (2.121) | 27 (2.236)

ADVERSE EVENTS:
Arm/Group | Intervention INVOS Cerebral Oximetry Monitoring | Standard of Care
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention INVOS Cerebral Oximetry Monitoring (N=12) | Standard of Care (N=13)
Death (Cardiac disorders) | 1 | 0 — Patient died during surgery as a result of aortic tear. Not related to study intervention.

LIMITATIONS AND CAVEATS:
The study was discontinued after 25 subjects completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes